CLINICAL TRIAL: NCT04657328
Title: Contrast-enhanced Ultrasound in Breast Tumor by Sonazoid
Brief Title: Prospective Multicenter Study on Clinical Application of Sonazoid in Breast Tumor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: S2020-300
Record Dates: First submitted 2020-09-26; First posted 2020-12-08 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Ultrasound
Keywords: breast

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — CNB in breast tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sonazoid as a new generation of ultrasound contrast agent.This study based on the features of Sonazoid specific angiography and high mechanical index,the role of Sonazoid in the differential diagnosis of breast benign and malignant tumors was explored.

DETAILED DESCRIPTION:
This trial is a prospective, multi-center study.With pathology as the gold standard, based on quantitative and qualitative analysis, Sonazoid-CEUS was compared with MRI to explore the diagnostic efficacy (accuracy, sensitivity and specificity) of Sonazoid-CEUS for breast tumor in different pathological types.

Investigators will also record the parameter information of imaging examination, pathological type of pathological examination and immunohistochemical index.Contrast-enhanced ultrasound includes lesion location, initial peak tumor volume, 1-minute tumor volume, 2-minute tumor volume, and 5-minute tumor volume, as well as the time for contrast enhancement, contrast agent clearance, and contrast agent clearance.Whether there is no enhancement area in the lesion after contrast enhancement, shape after contrast enhancement, edge after contrast enhancement, order of enhancement, uniformity of enhancement, intensity enhancement, pattern of enhancement, clear boundary after contrast enhancement, aspect ratio after contrast enhancement, etc.The magnetic field strength of the equipment is planned to be recorded in the enhanced MRI information, the name of the MRI contrast agent, the lesion location, the size of the LESION, and the scanning performance are enhanced (lump-like enhancement, non-lump-like enhancement, point-like enhancement), time-signal intensity enhancement curve, DWI signal, ADC value, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Conventional ultrasonography suggested definite lesions in the breast;
2. In addition to conventional ultrasound, there is also enhanced MRI examination;
3. There are no contraindications for puncture biopsy, and pathological examination (cytology, histology) is planned to examine the patients with target lesions
4. Patients volunteered to participate in the study and signed informed consent.-

Exclusion Criteria:

1. Those who are known to be allergic to ultrasound contrast agents;
2. The subject has a history of allergy to eggs or egg products (i.e. skin rash, dyspnea, swelling of the mouth or throat, hypotension or shock, etc.)
3. Arteriovenous (left and right) shunt patients in the heart and lungs
4. Patients with serious heart disease or serious lung disease
5. Patients who are pregnant, possibly pregnant or lactating
6. Patients who cannot receive contrast agent MRI
7. In addition, the investigator or the patient that the investigator considers not suitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Conventional ultrasonography suggested definite lesions in the breast;
  2. In addition to conventional ultrasound, there is also enhanced nuclear magnetic examination;
  3. There are no contraindications for puncture biopsy, and pathological examination (cytology, histology) is planned to examine the patients with target lesions
  4. Patients volunteered to participate in the study and signed informed consent.
Sampling Method: Probability Sample
Enrollment: 181 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of contrast-enhanced ultrasound in breast tumor by Sonazoid. | 10 months
  Pathology as a gold standard,to evaluate the diagnostic performance in breast tumor by Sonazoid.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lang M, Liang P, Shen H, Li H, Yang N, Chen B, Chen Y, Ding H, Yang W, Ji X, Zhou P, Cui L, Wang J, Xu W, Ye X, Liu Z, Yang Y, Wei T, Wang H, Yan Y, Wu C, Wu Y, Shi J, Wang Y, Fang X, Li R, Yu J. Head-to-head comparison of perfluorobutane contrast-enhanced US and multiparametric MRI for breast cancer: a prospective, multicenter study. Breast Cancer Res. 2023 May 30;25(1):61. doi: 10.1186/s13058-023-01650-3. PMID 37254149